CLINICAL TRIAL: NCT00317161
Title: Study to Show Lot-to-lot Consistency of Hib-MenAC Mixed With Tritanrix™-HBV, Its Non-inferiority to Tritanrix™-HBV/Hiberix™ With or Without Meningitec™, and MenA Response in 2, 4, 6 Month Infants With Hepatitis B Birth Dose
Brief Title: Immunogenicity & Safety Study of a Vaccine Against Meningitis in Infants (2,4,6 Months) After a Hepatitis B Birth Dose.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 100480
Record Dates: First submitted 2006-02-15; First posted 2006-04-24 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Hepatitis B; Haemophilus Influenzae Type b; Whole Cell Pertussis; Tetanus
MeSH Terms: conditions — Diphtheria; Hepatitis B; Haemophilus Infections; Tetanus

INTERVENTIONS:
Biological: DTPw-HBV/Hib-MenAC conjugate vaccine

SUMMARY:
The purpose of the study is to demonstrate consistent results in 3 production lots of Hib-MenAC vaccine when extemporaneously mixed with Tritanrix™-HepB and administered as a single injection, with respect to immunogenicity, safety and reactogenicity. Tritanrix™-HepB/Hiberix™ given alone and Wyeth Lederle's meningococcal C conjugate vaccine (Meningitec™), given concomitantly with Tritanrix™-HepB/Hiberix™ will be used as benchmark vaccines for all antigens except for MenA. The immunogenicity of MenA will also be evaluated.

DETAILED DESCRIPTION:
Randomized study with five groups to receive one of the following vaccination regimens after a birth dose of hepatitis B vaccine: One of the 3 lots of GSK Biologicals' Hib-MenAC mixed with GSK Biologicals' Tritanrix™-HBV (3 different groups) GSK Biologicals' Tritanrix™-HBV/Hiberix™ GSK Biologicals' Tritanrix™-HBV/Hiberix™ +Meningitec™

ELIGIBILITY:
Inclusion criteria:

• Healthy infants 56-83 days of age, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks and received a birth dose of hepatitis B vaccine within the first 72 hours of life.

Exclusion criteria:

* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history & physical examination.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine, or planned administration during the study period with the exception of oral polio vaccine (OPV).
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (>14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type b, and/or meningococcal disease.

Ages: 56 Days to 83 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2004-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Post-dose 3, bactericidal titers & antibody levels to meningococcal serogroups A & C; & PRP; & antibody levels to HBs, diphtheria, tetanus & BPT (subset of subjects).

SECONDARY OUTCOMES:
Solicited events (day 0-3); unsolicited events (day 0-30); serious adverse events (entire study). Pre-dose 1, antibody levels to Men(A&C) & PRP; & in some subjects anti-BPT antibody levels Seropositivity/seroprotection/vaccine response & antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kerdpanich A, Warachit B, Kosuwon P, Gatchalian SR, Watanaveeradej V, Borkird T, Kosalaraksa P, Han HH, Hutagalung Y, Boutriau D, Dobbelaere K. Primary vaccination with a new heptavalent DTPw-HBV/Hib-Neisseria meningitidis serogroups A and C combined vaccine is well tolerated. Int J Infect Dis. 2008 Jan;12(1):88-97. doi: 10.1016/j.ijid.2007.06.002. Epub 2007 Aug 22. PMID 17716936
- See also: Booster studies — http://www.clinicaltrials.gov/ct/show/NCT00136604
- Available data/document: Individual Participant Data Set: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register